CLINICAL TRIAL: NCT04697173
Title: Bundle Consent and Expectation Setting in Pediatric Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HM20019583
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Results first posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-03

CONDITIONS: Stress
MeSH Terms: interventions — Consent Forms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard consent (No Intervention): This group will be consented for invasive procedures using standard Hospital policy. Informed consent will be obtained either in person or via telephone with a witness from the patient or his/her legal guardian for any/all procedures medically indicated at that time, at the discretion of the Attending Physician.
- Bundled consent (Experimental): Upon admission, this group will received the document titled "Common PICU Procedures Explained" and encourage to read the document. They will then, within 24 hours of admission be consented using the Bundle Consent Document for the group of invasive procedures listed and explained in that document.
  Interventions: Other: Single consent

INTERVENTIONS:
Other: Single consent — A single consent form for possible procedures the child may undergo while in the PICU
  Arms: Bundled consent

SUMMARY:
The purpose of this research study is to find out about how obtaining consent for procedures in the PICU affects parental/caregiver stress. The researchers think that alleviating some of the uncertainly of a PICU stay by discussing types of procedural support offered and obtaining informed consent prior to their immediate necessity may help decrease stress experienced by caregivers. This study will allow the researchers to learn more about it.

DETAILED DESCRIPTION:
Having a child admitted to the Pediatric Intensive Care Unit (PICU) is a deeply challenging and stressful experience for parents and caregivers. Despite the high survival when compared to adult ICUs, a PICU admission can have meaningful long-term, negative health consequences for adult caregivers including symptoms of depression, anxiety and PTSD. There is little known in regards to what specific factors impact the mental health of parents/caregivers of PICU patients. However, research into stress and anxiety has suggested that uncertainty is a significant contributor to stress when faced with a new environment.

Usual informed consent for procedures performed in the PICU is obtained immediately prior to the procedure. Participants will be randomly assigned (like the flip of a coin) to either usual informed consent prior to each procedure or to a single consent form obtained upon admission to PICU for possible procedures their child may undergo. In this study participants will be asked to complete a survey at two separate times during the child's PICU hospitalization- 48-72 hours after admission and again upon transfer or discharge from the PICU. Data will be collected about the child from the medical record including age, diagnosis/reason for PICU admission, length of stay, and any procedures performed in PICU requiring consent.

ELIGIBILITY:
Inclusion Criteria:

* Parents/caregivers (>18 years) of children admitted to the Pediatric ICU during the designated study period

Exclusion Criteria:

* Anticipated length of PICU stay < 24 hours
* Non-English speaking parents/caregivers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nikki Miller Ferguson, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Society of Critical Care Medicine, Critical Care Statistics. Society of Critical Care Medicine, https://www.sccm.org/Communications/Critical-Care-Statistics. Retrieved 2020.
- [Background] Rodriguez-Rey R, Alonso-Tapia J, Colville G. Prediction of parental posttraumatic stress, anxiety and depression after a child's critical hospitalization. J Crit Care. 2018 Jun;45:149-155. doi: 10.1016/j.jcrc.2018.02.006. Epub 2018 Feb 16. PMID 29477091
- [Background] Durette, M. (2013). Uncertainty and Primary Appraisal as Predictors of Acute Stress Uncertainty and Primary Appraisal as Predictors of Acute Stress Disorder in Parents of Critically Ill Children: A Mediational Model. (Doctoral Thesis)
- [Background] Butler A, Copnell B, Willetts G. Family-centred care in the paediatric intensive care unit: an integrative review of the literature. J Clin Nurs. 2014 Aug;23(15-16):2086-99. doi: 10.1111/jocn.12498. Epub 2013 Dec 26. PMID 24372988
- [Background] Gill, M. PICU Prometheus: Ethical issues in the treatment of very sick children in Paediatric Intensive Care. Mortality, November 2005; 10(4): 262-275
- [Derived] Goldstein G, Karam O, Miller Ferguson N. The Effects of Expectation Setting and Bundle Consent on Acute Caregiver Stress in the PICU: A Randomized Controlled Trial. Pediatr Crit Care Med. 2023 Aug 1;24(8):692-700. doi: 10.1097/PCC.0000000000003265. Epub 2023 May 1. PMID 37125809

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study only enrolled parents/caregivers of children admitted to the pediatric ICU and the protocol enrollment reflects the number of parent participants.
Groups:
- Bundled Consent: Upon admission, this group will received the document titled "Common PICU Procedures Explained" and encourage to read the document. They will then, within 12 hours of admission be consented using the Bundle Consent Document for the group of invasive procedures listed and explained in that document.
  Single consent: A single consent form for possible procedures the child may undergo while in the PICU
Period: Overall Study
Arm/Group | Standard Consent | Bundled Consent
Started | 166 | 167
Completed | 132 | 129
Not Completed | 34 | 38
Not completed — Withdrawal by Subject | 34 | 38

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Consent | Bundled Consent | Total
Number analyzed (Participants) | 132 | 129 | 261
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 132 | 129 | 261
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 64 | 80 | 144
  Male | 66 | 48 | 114
  Did not identify | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 37 | 43 | 80
  White | 75 | 75 | 150
  More than one race | 9 | 4 | 13
  Unknown or Not Reported | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 132 | 129 | 261

OUTCOME MEASURES:

1. Primary Outcome: Parent/Caregiver Stress 48 to 72 Hours Following Admission to the Pediatric ICU
Description: Stress will be assessed using the Short Stress Overload Scale (SOS-S). The SOS-S is a 10 item questionnaire. Items are rated not at all (1) to a lot (5). Ratings are assigned a score and the scores are summed. Summed scores range from 10 - 50 with higher scores indicating greater stress. The SOS-S generates two subscores, Personal Vulnerability (PV) and Event Load (EL), with a score range from 5 to 25 for each. An individual's PV score corresponds to that individual's readiness to take on new stressors. Parents may be asked to complete the questionnaire multiple times depending on how long their child is in the PICU. This outcome measure only represents the PV portion of the SOS scale making the range from 5-25 (total of 5 questions each with a 1-5 scale).
Time Frame: 48 - 72 hours after admission of child to PICU
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard Consent | Bundled Consent
Number analyzed (Participants) | 132 | 129
units on a scale | 9 [5 to 14] | 8 [6 to 12]

2. Secondary Outcome: Number of Procedures Performed Without Appropriately Documented Consent
Description: Number of procedures preformed without recorded consent will be determined by reviewing child's medical chart. Stress will be assessed using the Short Stress Overload Scale (SOS-S). The SOS-S is a 10 item questionnaire. Items are rated not at all (1) to a lot (5). Ratings are assigned a score and the scores are summed. Summed scores range from 10 - 50 with higher scores indicating greater stress. The SOS-S generates two subscores, Personal Vulnerability (PV) and Event Load (EL), with a score range from 5 to 25 for each. An individual's EL score quantifies the stress burden placed on that individual by their current circumstances. Parents may be asked to complete the questionnaire multiple times depending on how long their child is in the PICU. This outcome measure only represents the EL portion of the SOS scale making the range from 5-25 (total of 5 questions each with a 1-5 scale).
Time Frame: At discharge or transfer out of PICU or 30 days after admission to the PICU, whichever comes first.
Measure: Mean (Inter-Quartile Range); unit: procedures
Arm/Group | Standard Consent | Bundled Consent
Number analyzed (Participants) | 132 | 129
procedures | 11 [6 to 15] | 9 [6 to 14]

3. Secondary Outcome: Parent/Caregiver Stress at Time of Discharge From the Pediatric ICU
Description: This was assessed by asking parent/caregiver a single question: "How life threatening do you believe your child's illness to be?" The question could be answered 1-5 with 1= not at all and 5= extremely.
Time Frame: At discharge or transfer out of PICU or 30 days after admission to the PICU, whichever comes first.
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard Consent | Bundled Consent
Number analyzed (Participants) | 132 | 129
units on a scale | 3 [2 to 5] | 3 [2 to 4]

ADVERSE EVENTS:
Time Frame: Up to 30 days
Arm/Group | Standard Consent | Bundled Consent
All-Cause Mortality (participants affected / at risk) | 4/132 | 3/129
Serious Adverse Events (participants affected / at risk) | 0/132 | 0/129
Other Adverse Events (participants affected / at risk) | 0/132 | 0/129

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT04697173/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT04697173/ICF_001.pdf